CLINICAL TRIAL: NCT05186207
Title: Women's Hospital School of Medicine Zhejiang University
Brief Title: Establishment of Special Disease Cohort for RPLand Study of Impact Mechanism of Early Embryo Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20210298-R
Record Dates: First submitted 2021-11-19; First posted 2022-01-11 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Recurrent Pregnancy Loss; Cohort Sutdy; Early Embryo Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: those who need clinical intervention before or after pregnancy, the experts shall formulate a personalized treatment plan according to the international guidelines. Researchers wouldn't interfere with the expert diagnosis and treatment process. And they should be confirmed intrauterine pregnancy within the study period.
  Interventions: Other: abnormal pre-pregnancy test results that need clinical intervention
- control group: those who need not clinical intervention before or after pregnancy, pregnancy was prepared under the clinical and health care guidance provided by experts, and intrauterine pregnancy was confirmed within the study period.

INTERVENTIONS:
Other: abnormal pre-pregnancy test results that need clinical intervention — The patients who need clinical intervention before or after pregnancy were divided into observation group. Doctors will formulate a personalized treatment plan according to the international guidelines. Researchers wouldn't interfere with the expert diagnosis and treatment process.
  Groups: observation group

SUMMARY:
Recurrent pregnancy loss (RPL) is a refractory disease with diverse etiologies, complex pathogenesis and limited therapeutic options. Current tests and treatments lack uniform specifications. This study is a prospective clinical cohort study which intends to screen out meaningful examination items and reliable and effective treatment. The study content includes (1) tracking the re-pregnancy information of patients with initial inevitable abortion, comparing the clinical data and examination test results between patients with single abortion and RPL, and (2) comprehensively and systematically screening the patients with initial inevitable abortion, taking those without obvious abnormalities and those with a re-pregnancy into the control group and taking those with a re-pregnancy after abnormal findings were treated into the study group, recording the pregnancy and perinatal conditions of the two groups, comparing the pregnancy outcomes of the two groups, and analyzing the risk factors for RPL. The results of this study will establish a model of maternal and newborn risk assessment for first trimester medication use and provide strong evidence-based evidence to clarify the diagnosis and treatment processes of RPL.

DETAILED DESCRIPTION:
Objective: (1) to establish a prediction model of pregnancy outcome and apply it to clinical practice; (2) to standardize the diagnosis and treatment of RPL.

This study is an observational study. The investigators only collect the medical data of patients without any intervention in the diagnosis and treatment plan. The data collection is in the charge of specially-assigned members of the investigators. The investigators set a security password for the database. The data is collected from outpatient medical record system, inpatient medical record system and questionnaire. One investigator is responsible for inputting the data into the database, and another investigator is responsible for checking the Corrigendum.

1. Before enrollment, the investigators would record the medical history of the couple in detail, including age, menstruation, marriage and reproductive history, family history, and the details of previous abortion.
2. The following examinations should be completed before pregnancy: in addition to the routine pre-pregnancy examination items, the examination items related to recurrent spontaneous abortion were added, including uterine artery resistance ultrasound, couple's chromosome, reproductive hormone, OGTT test and some immune related indexes.
3. According to the examination results, the experts of recurrent spontaneous abortion team would evaluate the patients and divided them into:

1) Control group:those who needn't clinical intervention before or after pregnancy , pregnancy was prepared under the clinical and health care guidance provided by experts, and intrauterine pregnancy was confirmed within the study period.

2) Observation group: those who need clinical intervention before or after pregnancy, the experts shall formulate a personalized treatment plan according to the international guidelines. Investigators wouldn't interfere with the expert diagnosis and treatment process. And they should be confirmed intrauterine pregnancy within the study period.

(4) The investigators monitored and tracked the indicators during pregnancy and perinatal period of the two groups, including:

1. The participants should complete the routine health care and necessary examination items on schedule, which is the same as that of normal pregnant women.
2. Coagulation function and immune function related tests will be performed respectively in early pregnancy, middle pregnancy and late pregnancy respectively.
3. Length of cervical canal will be check at least once in the second trimester of pregnancy. Uterine artery blood flow was monitored by ultrasound at least every 4 weeks from early pregnancy until 24 weeks of pregnancy. The fetal growth measurement ultrasound was performed respectively at 20 weeks, 28 weeks, 32 weeks and 36 weeks of gestation.
4. Additional OGTT test at 12-16 weeks of gestation.
5. Tests of glucose and lipid metabolism indexes of maternal blood and urine during early, middle and late pregnancy.

(5) When the participant is hospitalized for delivery, the investigators will collect the following data: length of hospital stay, diagnosis, fetal position, number of pregnancies, weight gain before delivery, mode of delivery, postpartum hemorrhage, puerperal infection, neonatal birth weight, neonatal Apgar score and examination results during and after delivery.

(6) The following analysis shall be made according to the obtained medical data:

1. The statistical differences of various indexes between the two groups were compared.
2. The abortion rate, preterm birth rate and other pregnancy outcomes were compared between the two groups.
3. Multivariate analysis was used to analyze the independent risk factors of recurrent abortion.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients who were treated in the outpatient department of Zhejiang University Women's Hospital from January 1, 2018 to December 31, 2020;
* (2) With history of once spontaneous abortion;
* (3) Having fertility requirements but not yet pregnant;
* (4) Those who are willing to give birth again during the study period.

Exclusion Criteria:

* (1) Previous history of multiple spontaneous abortion, inevitable abortion or missed abortion;
* (2) Re pregnancy after abortion, now in pregnancy or delivered;
* (3) Patients who are participating in other clinical studies or those who refuse to participate in the study;
* (4) The researchers consider that she is not suitable to participate in this study for other reasons.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who were treated in the outpatient department of Zhejiang University Women's Hospital from January 1, 2018 to December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-12 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with different pregnant outcome | From date of enrollment until the date of termination of pregnancy, assessed up to 24 months.
  Number of participants with abortion, preterm birth, stillbirth, induced labor, flat birth or cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China